CLINICAL TRIAL: NCT05428189
Title: Efficacy of the Disclosing Plaque Agent as a Guide to Remove the Oral Biofilm in Orthodontic Patients: a Randomised Controlled Trial Study
Brief Title: Efficacy of the Disclosing Plaque Agent as a Guide to Remove the Oral Biofilm in Orthodontic Patients.
Acronym: ORTOPLAK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Magda Mensi, Principal investigator, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ORTOPLAK
Record Dates: First submitted 2022-06-08; First posted 2022-06-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Plaque
Keywords: Oral Hygiene; Dental Care; Orthodontic Patient; Disclosing Plaque Agent
MeSH Terms: conditions — Plaque, Amyloid

STUDY DESIGN:
Intervention Model Description: Monocetric, single blinded, randomized clinical trial, parallel design.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided Biofilm Therapy (GBT) (Experimental): The subjects receive professional oral hygiene guided by plaque a disclosing agent, using air-polishing and a ultrasonic device
  Interventions: Diagnostic Test: Plaque Disclosing Agent; Device: Airpolishing and ultrasonic debridement
- Air Polishing and Ultrasonic Debridment (Active Comparator): The subject receive professional oral hygiene using air-polishing and a ultrasonic device
  Interventions: Device: Airpolishing and ultrasonic debridement

INTERVENTIONS:
Diagnostic Test: Plaque Disclosing Agent — A plaque disclosing agent is applied on teeth to detect plaque. Air-polishing will be used as main instrument for biofilm and stains removal, followed by ultrasonic scaling.
  Arms: Guided Biofilm Therapy (GBT)
Device: Airpolishing and ultrasonic debridement — Air-polishing will be used as main instrument for biofilm and stains removal, followed by ultrasonic scaling.

SUMMARY:
It is more difficult to perform excellent professional oral hygiene in patients wearing orthodontic appliances.

The hypothesis of the present randomized controlled trial is that the application of plaque disclosing agent allows better biofilm removal.

To test this hypothesis, the patients, upon initial evaluation, will be divided in 2 study groups:

* CONTROL GROUP will receive professional oral hygiene without disclosing agent
* TEST GROUP will receive professional oral hygiene guided by plaque disclosing agent

At the end of the professional oral hygiene session, the disclosing agent is re-applied in all patients and the percentage of residual plaque area is calculated though image software analysis (ImageJ).

DETAILED DESCRIPTION:
Oral biofilm is not always visible, so its complete removal can be challenging. Applying a plaque disclosing agent before the therapy might serve as a guide to better remove biofilm. Thanks to this tool, the clinicians can clearly see where the plaque is, so its removal can be more thorough.

In orthodontic patients, it is even more difficult to remove biofilm and plaque, as the fixed appliances pose an obstacle. The hypothesis is that using a plaque disclosing agent as a guide to the operator, better removal of the biofilm can be achieved.

The study will be performed to assess the efficacy of disclosing plaque agent as a guide to remove biofilm and plaque in orthodontic patients during professional oral hygiene, performed with air-polishing with erythritol powder and a ultrasonic device.

TRIAL DESIGN: Monocetric, pragmatic, single blinded, randomized clinical trial (RCT) of parallel design.The trial will have one-year duration.

STUDY POPULATION: Orthodontic patients with plaque index above the 25% and without periodontal disease.

PRIMARY OUTCOME: the percentage of area in which the disclosing plaque agent is present after the treatment (RPA: Residual Plaque Area).

RPA: residual plaque area: percentage of area with residual plaque coloured by plaque disclosing agent. This will be analysed and calculated with a image analysis software (ImageJ).

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form;
* Male and female subjects, aged 18-75 years, inclusive;
* Presence of orthodontic appliances;
* Good general health (free of systemic diseases such as diabetes, HIV infection or genetic disorder, ongoing malignant disease of any type that could influence the outcome of the treatment and might interfere with the evaluation of the study objectives);
* Generalized gingivitis;
* Plaque index (PI) above 25%;
* Availability for session of the study for an assigned subject;
* Presence of all inferior and superior anterior teeth from canine to canine;
* Smoking less than 10 cigarettes a day.

Exclusion Criteria:

* Chronic obstructive pulmonary disease and asthma;
* Patients with periodontally disease defined as presence of PPD >= 4mm and /or PAL of >=3m;
* Splinted teeth;
* Presence of prosthesis;
* Tumors or significant pathology of the soft or hard tissues of the oral cavity;
* Current radiotherapy or chemotherapy;
* Pregnant or lactating women;
* History of allergy to Erythritol;
* History of adverse reactions to lactose or fermented milk products;
* Restorations on the teeth to be treated which may interfere with treatment administration and/or scoring procedures, at the discretion of the examiner;
* Not willing to follow the agreed protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-10-10 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Residual Plaque Area (RPA) | At the end of the treatment session
  The percentage of area in which plaque is still present, as revealed by re-application of plaque disclosing agent, in both groups at the end of the treatment session

CONTACTS AND LOCATIONS:
Overall Officials: Magda Mensi, Principal Investigator — ASST Spedali Civili di Brescia
Locations (1):
- Magda, Brescia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-29): https://cdn.clinicaltrials.gov/large-docs/89/NCT05428189/Prot_SAP_000.pdf